CLINICAL TRIAL: NCT07068503
Title: Running Injuries, Patient-Specific Quality of Life, Injury Prevention and Treatment Habits Among the Romanian-Speaking Population
Brief Title: Study of Running Injuries and Treatment Habits in Romanian Speakers
Status: Not yet recruiting | Type: Observational
Sponsor: University of Pecs (Other)
Responsible Party: Sponsor
Other Study IDs: 8393/ 3/ 10.06.2024
Record Dates: First submitted 2025-06-25; First posted 2025-07-16 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-06

CONDITIONS: Running; Health Care Seeking Behavior; Manual Therapies; Health Surveys; Running Related Injuries; Validation Studies; Surveys and Questionnaires
Keywords: Health Behavior; Health Care Seeking Behavior; Running; Running related injury; Cross-Sectional Studies; Treatment Habits; Romanian Population; Sports Medicine; Healthcare Utilization; Manual therapies; Quality of Life; Questionnaire Validation; UWRI
MeSH Terms: conditions — Patient Acceptance of Health Care; Health Behavior

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study examines running injuries, quality of life, and treatment habits among Romanian-speaking runners. A key objective is the Romanian language adaptation and validation of the University of Wisconsin Running Injury and Recovery Index (UWRI), a running-specific questionnaire.

The purpose is to understand:

* What types of running injuries are most common
* How injuries affect runners' daily life and well-being
* What prevention and treatment methods runners currently use
* What healthcare services runners use for injuries
* To provide a validated Romanian version of the UWRI questionnaire

Participants will complete an online questionnaire about their running experience, any injuries they have had, how these injuries affected their life, and what treatments they tried.

The survey takes about 25-30 minutes to complete. All information is confidential and anonymous.

This research will help healthcare providers better understand and treat running injuries in the Romanian-speaking community.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Romanian native speakers
* Recreational or competitive runners defined as individuals who have been running for at least 1 year prior to questionnaire completion with minimum 5 km per week
* Voluntary participation and willing to provide informed consent

Exclusion Criteria:

* Lower extremity traumatic injuries not related to running (fractures, dislocations, etc.)
* Neurological diseases with muscle weakness
* Rheumatoid arthritis affecting lower extremities
* Irregular runners who do not meet the minimum running criteria
* Under 18 years of age
* Non-Romanian native speakers
* Unwilling to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Romanian-speaking running community members recruited through online running groups, social media platforms, and running clubs across Romania. Participants will be identified through purposive sampling from recreational and competitive running communities.
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2025-07-30 (Estimated); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Reliability and Validity of Romanian Running Injury Questionnaire | Baseline
  Assessment of psychometric properties of the Romanian version of University of Wisconsin Running Injury and Recovery Index (UWRI), a questionnaire that measures running injuries and recovery. The UWRI scale ranges from 0 to 36, where higher scores indicate greater running ability. Reliability measured using Cronbach's alpha coefficient for internal consistency. Validity assessed through factor analysis and correlation with quality of life measures. Cronbach's alpha ranges from 0 to 1, where 0 indicates no reliability and 1 indicates perfect reliability. Values above 0.70 indicate acceptable reliability, above 0.80 indicate good reliability.

SECONDARY OUTCOMES:
Healthcare Utilization Patterns for Running Injuries | Baseline
  Proportion of participants who consulted healthcare providers for running-related injuries, assessed through structured questionnaire. Categorized by provider type (physicians, physiotherapists, sports medicine specialists), frequency of visits and types of treatments received. Healthcare-seeking behavior patterns will be reported as percentages and frequencies among Romanian runners with injuries.
Manual Therapy Knowledge and Attitudes Assessment for Running Injuries | Baseline
  Assessment of knowledge, attitudes, and utilization patterns regarding manual therapy among runners using structured questionnaire. Includes perceived effectiveness, awareness of benefits, previous utilization, and willingness to seek manual therapy treatment. Results reported as descriptive statistics and categorical responses.